CLINICAL TRIAL: NCT07325942
Title: Effectiveness of Low -Versus High -Volume High -Intensity Interval Training in Patients With Chronic Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Ibrahim Elshenawy Elshenawy, physical therapy specialist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005825
Record Dates: First submitted 2025-12-09; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low volume high intensity interval training (Experimental): This group will receive the usual care (standard medical treatment) in addition to LV-HIIT on a treadmill for 8 weeks, 2 sessions per week.
  Interventions: Other: low-volume high intensity interval training; Drug: Standard medical treatment
- high volume high intensity interval training (Experimental): In this group, the patients will receive the usual care (standard treatment) in addition to HV-HIIT on a treadmill for 8 weeks, 2 sessions per week
  Interventions: Other: High volume high intensity interval training; Drug: Standard medical treatment
- control group (Other): It includes 15 patients who will receive standard medical treatment only
  Interventions: Drug: Standard medical treatment

INTERVENTIONS:
Other: low-volume high intensity interval training — Low-volume HIIT (LV-HIIT) is a particularly time-efficient subtype of interval training, which has gained increasing attention in recent years. As per the previous definition, these brief training protocols typically involve≤10 min of intense exercise within a session lasting≤30 min including warm-up, recovery phases between intervals, and cool-down
  Arms: Low volume high intensity interval training
Other: High volume high intensity interval training — long (2-4 min) bouts of high (not maximum) intensity exercise interspersed with recovery periods which have wide varieties in the protocols according to the intensity, duration, and number of intervals performed
  Arms: high volume high intensity interval training
Drug: Standard medical treatment — standard medical treatment for chronic heart failure as per international guidlines

SUMMARY:
this study aims to investigate the effect of low vs high volume- high intensity interval training on functional capacity and quality of life in chronic heart failure patients

ELIGIBILITY:
Inclusion Criteria:

1. Chronic stable heart failure patient with reduced ejection fraction (EF <40)
2. Age Above 18 years old
3. Both males and females
4. The ability to provide informed consent

Exclusion Criteria:

1. Based on the Scientific Statement from the American Heart Association: contraindications for exercise Testing and Training. (Fletcher et al., 2013)

   1. Acute myocardial infarction (MI), within 2 days
   2. Ongoing unstable angina
   3. Uncontrolled cardiac tachy or brady arrhythmia with hemodynamic compromise
   4. Active endocarditis
   5. Symptomatic severe aortic stenosis
   6. Decompensated heart failure
   7. Acute pulmonary embolism, pulmonary infarction, or deep vein thrombosis
   8. Acute myocarditis or pericarditis
   9. Acute aortic dissection
   10. Physical disability that precludes safe and adequate testing or training
   11. Known obstructive left main coronary artery stenosis
   12. Hypertrophic obstructive cardiomyopathy with severe resting gradient
   13. Recent stroke or transient ischemic attack
   14. Mental impairment with limited ability to cooperate
   15. Resting hypertension with systolic or diastolic blood pressures >200/110 mmHg
   16. Uncorrected medical conditions, such as significant anemia, important electrolyte imbalance, and hyperthyroidism
2. Acute decompensated heart failure NYHA class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-06-06 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
6 minute walk test | at enrolment and at the end of treatment at 8 weeks
  self-paced submaximal field exercise test to assess submaximal functional capacity of the patient , the distance walked by the patient for six minutes will be measured by meters
2D Echocardiographic parameters | at enrollment and at the end of treatment at 8 weeks
  Left ventricle geometry: left ventricular end-diastolic diameter (LVEDD) mm, left ventricular end-systolic diameter (LVESD) mm, left ventricular end-systolic volume (LVESV) ml. and, left ventricular end-diastolic volume (LVEDV) ml.
  Left ventricle Systolic function: left ventricular ejection fraction (LVEF) % Left ventricle Diastolic function :E wave cm/s: early diastolic mitral inflow velocity, A wave cm/s: diastolic mitral inflow velocity during late atrial contraction , E/A ratio

SECONDARY OUTCOMES:
Minnesota living with heart failure questionnaire (MLHFQ) | at enrollment and at the end of treatment at 8 weeks
  The Minnesota Living with Heart Failure Questionnaire (MLHFQ) is the tool most widely used and recognized to assess HRQOL in adults with Hf, was developed in 1987 by Thomas Rector, focusing on the underlying relationship between pathophysiology, symptoms, functional limitations, and psychological distress, it measures the impacts of symptoms and treatment on different dimensions of HRQOL in HF patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt